CLINICAL TRIAL: NCT05191303
Title: Developing Mobile Intervention of the Breast Feeding Counseling and Evaluating Its Effectiveness in Primiparous Mothers
Brief Title: Effectiveness of Mobile Intervention for Breast Feeding Counseling (MIBFc) in Primiparous Mothers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oulu (Other)
Collaborators: Oulu University Hospital (Other)
Responsible Party: Principal Investigator, Pirkko Nikula, Principal Investigator, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1954032
Record Dates: First submitted 2021-12-10; First posted 2022-01-13 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Breast Feeding, Exclusive
Keywords: Mobile application; Attitude; Confidence, Self; Counseling; Intervention; Randomized controlled trial (RCT); Breast Feeding, exclusive; Primiparous
MeSH Terms: conditions — Breast Feeding; Behavior

STUDY DESIGN:
Intervention Model Description: A single-blind randomized controlled trial with a two-arm design will be conducted among primiparous mothers. Participants are randomized to two groups, a intervention and a control group. Participants receive standard usual care of breastfeeding counselling in both groups. In addition, the intervention group members will use mobile intervention of breastfeeding counseling.
Who Masked: Participant
Masking Description: Statistician, who is not involved in the study has done block-randomization with variable block-sizes (2,4,6) by StatsDirect program for two groups; an intervention and control group. Maternity care staff asks informed consent and then performs the randomization of primiparous women to the intervention or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): In addition to standard usual care of breastfeeding counseling, the intervention group will have an opportunity to access the mobile application breastfeeding counseling from weeks 18 of pregnancy, continuing for up to 6 months after childbirth.
  Interventions: Device: Mobile intervention of breastfeeding counseling
- Control group (No Intervention): The control group receives the standard usual care of breastfeeding counseling in maternity care and in hospital from weeks 18 of pregnancy, continuing for up to 6 months after childbirth.
  The standard usual care of breastfeeding follows the 10 steps of the Baby Friendly Hospital Initiative programme and Finnish Institute for Health and Welfare recommendation.

INTERVENTIONS:
Device: Mobile intervention of breastfeeding counseling — The mobile intervention of breastfeeding counseling includes an evidence-based information of breastfeeding, which is based on Ten steps of breastfeeding of Baby Friendly Hospital Initiative (BFHI) and Finnish Institute for Health and Welfare recommendation. The links provide more information and videos related to breastfeeding topic. The mobile intervention of breastfeeding counseling allows the client to write comments or notes that can be used in counseling at maternity clinic or hospital. The mobile intervention of breastfeeding counseling also provides an e-mail to non-urgent questions related to breastfeeding. Questions will be answered within 3 or 4 days by a lactation consultant (IBCLC).
  Arms: Intervention group

SUMMARY:
The purpose of this study is to evaluate the effectiveness of mobile intervention for breastfeeding counseling (MIBFc) to improve exclusive breastfeeding duration among primiparous women in Finland.

DETAILED DESCRIPTION:
The investigators hypothesize that the use of mobile intervention for breastfeeding counseling to primiparous women improve the exclusive breastfeeding rates, breastfeeding attitudes, breastfeeding confidence and the satisfaction of breastfeeding counselling. These outcomes are assumed to be higher in the intervention group than in the control group.

ELIGIBILITY:
Inclusion Criteria:

* primiparous women
* 18 years or older
* finnish language
* singleton foetus
* have an intention to breastfeed
* have a smartphone

Exclusion Criteria:

* multiple pregnancy
* risk pregnancy, or other disease to be monitored

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 228 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Exclusive breastfeeding relative rate at 1 months of age | 1 month after childbirth
  Proportion of infants exclusive breastfeeding at 1 month: Exclusive breastfeeding is defined when the infant only receives breast milk, D-vitamin and needed medicines.
Exclusive breastfeeding relative rate at 4 months of age | 4 moths after childbirth
  Proportion of infants exclusive breastfeeding at 4 month: Exclusive breastfeeding is defined when the infant only receives breast milk, D-vitamin and needed medicines.
Exclusive breastfeeding relative rate at 6 months of age | 6 months after childbirth
  Proportion of infants exclusive breastfeeding at 6 month: Exclusive breastfeeding is defined when the infant only receives breast milk, D-vitamin and needed medicines.

SECONDARY OUTCOMES:
The Iowa Infant Feeding Attitude Scale (IIFAS) at pregnancy | Measurements are made in 18 and 34 weeks of gestation
  IIFAS is a 17-items scale developed by De la Mora and Russell (1999) to evaluate maternal attitudes toward infant feeding. The Scale relatively easy to administer and score and it is usable with a wide variety of populations. Scale is 5 point Likert type scale.
Breastfeeding Self-Efficacy Scale- Short Form (BSES-SF) | Measurements are made in 1 and 4 months after childbirth
  Breastfeeding Self-Efficacy Scale-Short Form: It is a 33-item scale developed by Dennis and Faux (1999) to evaluate breastfeeding self-efficacy levels of mothers. Later, a 14-item short form of the scale was developed in 2003 (Dennis 2003). Dennis (2003) recommends this short form for use. It is applied more easily and evaluates self-efficacy correctly. Breastfeeding Self-Efficacy Short Form Scale is a 5 point Likert type scale.
Satisfaction of breastfeeding guidance | Measurements are made in 18 and 34 weeks of gestation, and in 1 and 4 months after childbirth.
  Satisfaction of breastfeeding guidance measured with Visual Analogue Scale (VAS) (numeric 0 to 10)
Use of infants additional milk at hospital after childbirth | The researcher retrieves the data from the patient record after 6 months of childbirth.
  Use of infants additional milk at hospital after childbirth and only medical supplementary milk accepted
Infants exclusive breastfeeding rate (relative share / portion) | The researcher retrieves the data from the patient record after 6 months of childbirth.
  Infants exclusive breastfeeding rate (relative share / portion) when leaving the hospital. Only medical supplementary milk accepted

CONTACTS AND LOCATIONS:
Locations (1):
- City of Oulu Maternity Clinic, Oulu, Finland